CLINICAL TRIAL: NCT00001813
Title: Examination of Clinical and Laboratory Abnormalities in Patients With Defective DNA Repair: Xeroderma Pigmentosum, Cockayne Syndrome, or Trichothiodystrophy
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990099; 99-C-0099; NCT00004044 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-06-13

CONDITIONS: Cockayne Syndrome; Skin Neoplasms; Xeroderma Pigmentosum; Trichothiodystrophy Syndromes; Genodermatosis
Keywords: Xeroderma Pigmentosum; Trichothiodystrophy; Cockayne Syndrome; Skin Cancer; DNA Repair; Natural History
MeSH Terms: conditions — Cockayne Syndrome; Skin Neoplasms; Xeroderma Pigmentosum; Trichothiodystrophy Syndromes; Skin Diseases, Genetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Subjects with clinical and/or laboratory documentation of typical features or suggestiveclinical features of XP, CS, TTD, or overlap syndromes
- 2: Family members of patients with XP, CS, TTD, or overlap syndromes
- 3: Healthy volunteers

SUMMARY:
Four rare genetic diseases, xeroderma pigmentosum (XP), Cockayne syndrome (CS), the XP/CS complex and trichothiodystrophy (TTD) have defective DNA excision repair although only XP has increased cancer susceptibility. We plan to perform careful clinical examination of selected patients with XP, XP/CS, CS, or TTD and follow their clinical course. We will obtain tissue (skin, blood, hair, buccal swabs) for laboratory examination of DNA repair and for genetic analysis. We hope to be able to correlate these laboratory abnormalities with the clinical features to better understand the mechanism of cancer prevention by DNA repair. Patients will be offered counseling and education for cancer control....

DETAILED DESCRIPTION:
Three rare genetic diseases, xeroderma pigmentosum (XP), Cockayne syndrome (CS), and trichothiodystrophy (TTD) have defective DNA excision repair although only XP has increased cancer susceptibility. We plan to perform careful clinical examination of selected patients with XP, CS, TTD, or overlap syndromes to follow their clinical course. We will obtain tissue (skin, blood, hair, or buccal cells) for laboratory examination of DNA repair and for histologic, protein, biochemical, and genetic analysis. We hope to be able to correlate these laboratory abnormalities with the clinical features to better understand the mechanism of cancer prevention by DNA repair. Patients will be offered counseling and education for cancer control.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects age 6 weeks and above:

  * with clinical and/or laboratory documentation of typical features or suggestive clinical features of XP, CS, TTD, or overlap syndromes or
  * that are first degree relatives or other family members of participants with XP, CS, TTD, or overlap syndromes
* Healthy volunteers of age 1 year and above (including NIH employees) willing to donate blood, skin, buccal cells, or hair.
* Patients or legally authorized representatives must provide informed consent.

EXCLUSION CRITERIA:

-Inability or unwillingness to provide tissue (skin, blood, buccal cells or hair) for laboratory studies.

Ages: 6 Weeks to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be sought by contacting professional organizations (such as the American Academy of Dermatology-XP Task Force), lay support groups (such as the XP Society and the Share and Care CS Support Network) or by direct referral. Healthy volunteers or NIH staff will be recruited through the Program for Healthy Volunteers (CRVP@mail.cc.nih.gov), through the Patient Recruitment and Public Liaison Office (prpl@mail.cc.nih.gov), or as a self-referral through the clinicaltrials.gov web site (http://clinicaltrials.gov). Healthy volunteers may also be approached by a member of the LCBG, NCI regarding interest in participating on this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 709 (Actual)
Dates: Start 1999-05-10 (Actual)

PRIMARY OUTCOMES:
Identify patients with genetic diseases | Up to 3 days
  Proportion of patients with three rare genetic diseases; xeroderma pigmentosum (XP), Cockayne syndrome (CS), and trichothiodystrophy (TTD)and overlap syndromes

SECONDARY OUTCOMES:
Diagnosis confirmation | up to 3 days
  -To confirm suspected cases of XP, CS, TTD, XP/TTD or overlap syndrome patients by review of clinical records, by clinical examination and by laboratory testing -To document presence (or absence) of cancers (skin, eye, tongue, or internal) in XP, XP/CS, CS, TTD, XP/TTD and other overlap syndrome patients-To document atypical clinical features or unusual environmental exposures of patients with XP, XP/CS, CS, TTD, XP/TTD and otheroverlap syndromes
Tissue collection | up to 3 days
  obtain tissue (skin, blood, hair or buccal cells) from XP, CS, TTD, XP/TTD or overlap syndrome patients, their first-degree relatives and healthy volunteers for establishment of cell cultures and for examination of DNA repair and genetic analysis
identify molecular defects | up to 3 days
  identify molecular defects in the DNA repair or other genes in cells from patients with XP, CS, TTD, XP/TTD or overlap syndromes and toattempt to correlate the defects with the clinical features
overall survival | yearly
  follow the clinical course of selected patients with XP, CS, TTD, XP/TTD or overlap syndromes

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Sargen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: -Clinical data available during the study and indefinitely.@@@@@@-Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active
Access Criteria: -Clinical data will be made available and with the permission of the study PI.@@@@@@-Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Barrett SF, Robbins JH, Tarone RE, Kraemer KH. Evidence for defective repair of cyclobutane pyrimidine dimers with normal repair of other DNA photoproducts in a transcriptionally active gene transfected into Cockayne syndrome cells. Mutat Res. 1991 Nov;255(3):281-91. doi: 10.1016/0921-8777(91)90032-k. PMID 1719400
- [Background] Boltshauser E, Yalcinkaya C, Wichmann W, Reutter F, Prader A, Valavanis A. MRI in Cockayne syndrome type I. Neuroradiology. 1989;31(3):276-7. doi: 10.1007/BF00344359. PMID 2779780
- [Derived] Merideth M, Tamura D, Angra D, Khan SG, Ferrell J, Goldstein AM, DiGiovanna JJ, Kraemer KH. Reproductive Health in Xeroderma Pigmentosum: Features of Premature Aging. Obstet Gynecol. 2019 Oct;134(4):814-819. doi: 10.1097/AOG.0000000000003490. PMID 31503159
- [Derived] Atkinson EC, Thiara D, Tamura D, DiGiovanna JJ, Kraemer KH, Hadigan C. Growth and nutrition in children with trichothiodystrophy. J Pediatr Gastroenterol Nutr. 2014 Oct;59(4):458-64. doi: 10.1097/MPG.0000000000000458. PMID 24918982
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-C-0099.html